CLINICAL TRIAL: NCT04450238
Title: The Dual Factor Model of Mental Health: A Longitudinal Study in Inpatients
Brief Title: The Dual Factor Model of Mental Health in Inpatients
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Stillachhaus Privatklinik (Unknown)
Responsible Party: Principal Investigator, Ruth von Brachel, Principal Investigator, Ruhr University of Bochum
Other Study IDs: 2017-387
Record Dates: First submitted 2020-06-10; First posted 2020-06-29 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Psychological Disease; Depression
Keywords: Dual Factor Model; Positive mental health; Suicidal ideation
MeSH Terms: conditions — Depression; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: All participants are inpatients at the clinic "Stillachhaus" in Germany. They are receiving treatment for a variety of psychological disoders, mostly depressive disoders.
  Interventions: Behavioral: Routine care inpatient treatment

INTERVENTIONS:
Behavioral: Routine care inpatient treatment — All participants are receiving inpatient treatment consisting of a variety of psychological interventions such as cognitive-behavioral therapy, third-wave interventions, psycho-education and in some cases medication.

SUMMARY:
The Dual Factor Model of mental health (DFM; Greensporn & Saklofske, 2001) postulates that mental health consists of two at least partially unrelated factors, the experience or absence of psycho-pathological symptoms (i.e. depressive symptoms) and the experience or absence of positive mental health (i.e. life satisfaction, meaningfulness). Both factors contribute to an individual's well-being and mental health.The DFM has been used as a framework to describe and evaluate participants' mental health in different settings in cross-sectional and longitudinal designs mostly outside of clinical settings. Psychological Interventions, such as cognitive-behavioral therapy are widely studied concerning their reduction of psycho-pathological symptoms. However, little is known about the effect of psychological interventions on the second factor (positive mental health) of the DFM. This is especially important, because the latter has been shown to contribute significantly to subjective well-being and to reduce the risk of suicidal intentions and behavior.

Primary, the authors aim to investigate the DFM in an inpatient sample over the course of time (pre-treatment, post-treatment, 6 and 12 months after discharge). Secondly, they aim to investigate the relationship between positive mental health and suicidal ideation over the course of time.

DETAILED DESCRIPTION:
Participants will be divided into four groups according to the DFM over the course of time:

1. unhappy: high psychopathology and low positive mental health; depression and/or anxiety scores above published cut -offs and positive mental health scores under published cut offs.
2. symptomatic but content: high psychopathology and high positive mental health; depression and/or anxiety scores above published cut -offs and normal to high positive mental health scores
3. vulnerable: low psychopathology and low positive mental health; depression and/or anxiety scores under published cut -offs and positive mental health scores under published cut offs
4. Complete mental health: low psychopathology and high positive mental health; depression and/or anxiety scores under published cut -offs normal to high positive mental health scores.

The authors will then depict the movements of patients through these groups graphically and use regression analyses to check for differences according to age, diagnosis and gender.

Towards the second aim they will use regression analyses to investigate the protective effect of positive mental health on suicidal ideation or behavior.

ELIGIBILITY:
Inclusion Criteria:

-inpatients at the Stiilachaus Privatklinik

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients at Stillachhaus Privatklinik fill out the questionnaires prior and post treatment as part of their routine assessment. They are invited to fill out the same measures 6 and 12 months after discharge voluntarily to support the long-term evaluation of their treatment. They have all given written informed consent to use their data for publication.
Sampling Method: Probability Sample
Enrollment: 1552 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale-21 (DASS-21; Nilges et al., 2016) | In the first 3 days of treatment
  Measures depression, anxiety and stress with 21 items. Scores range from 0-63 with higher scores indicating more severe anxiety, depression and stress.
Depression Anxiety Stress Scale-21 (DASS-21; Nilges et al., 2016) | In the last three days of treatment
  Measures depression, anxiety and stress with 21 items. Scores range from 0-63 with higher scores indicating more severe anxiety, depression and stress.
Depression Anxiety Stress Scale-21 (DASS-21; Nilges et al., 2016) | 6 months after discharge
  Measures depression, anxiety and stress with 21 items. Scores range from 0-63 with higher scores indicating more severe anxiety, depression and stress.
Depression Anxiety Stress Scale-21 (DASS-21; Nilges et al., 2016) | 12 months after discharge
  Measures depression, anxiety and stress with 21 items. Scores range from 0-63 with higher scores indicating more severe anxiety, depression and stress.
Positive mental health scale (PMH; Lukat et al., 2016) | In the first 3 days of treatment
  Measures positive psychological functioning with 9 items. Scores range from 0-27 with higher scores indicating more positive mental health.
Positive mental health scale (PMH; Lukat et al., 2016) | In the last three days of treatment
  Measures positive psychological functioning with 9 items. Scores range from 0-27 with higher scores indicating more positive mental health
Positive mental health scale (PMH; Lukat et al., 2016) | 6 months discharge
  Measures positive psychological functioning with 9 items. Scores range from 0-27 with higher scores indicating more positive mental health
Positive mental health scale (PMH; Lukat et al., 2016) | 12 months discharge
  Measures positive psychological functioning with 9 items. Scores range from 0-27 with higher scores indicating more positive mental health.

SECONDARY OUTCOMES:
Suicidal Behavior Questionnaire (SBQ; Osman et al., 2001) ). | In the first 3 days of treatment
  Assesses past and current suicidal ideation and behavior. Scores range from 3-18 with higher scores indicating a higher risk for suicidal behavior.
Suicidal Behavior Questionnaire (SBQ; Osman et al., 2001) ). | In the last three days of treatment
  Assesses past and current suicidal ideation and behavior. Scores range from 3-18 with higher scores indicating a higher risk for suicidal behavior.
Suicidal Behavior Questionnaire (SBQ; Osman et al., 2001) ). | 6 months after discharge
  Assesses past and current suicidal ideation and behavior. Scores range from 3-18 with higher scores indicating a higher risk for suicidal behavior.
Suicidal Behavior Questionnaire (SBQ; Osman et al., 2001) ). | 12 months after discharge
  Assesses past and current suicidal ideation and behavior. Scores range from 3-18 with higher scores indicating a higher risk for suicidal behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Margraf, Prof., Study Director — Ruhr-University Bochum
Locations (1):
- Stillachhaus Privatklinik, Oberstdorf, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Since we do not have written consent to publish the data we will refrain from making it publicly available.